CLINICAL TRIAL: NCT02755948
Title: Cell Mediated Immunity Against RSV and Influenza in a Human Experimental Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13SM0365; 11/LO/1826 (Other: London-Fulham Research Ethics Committee)
Record Dates: First submitted 2016-04-11; First posted 2016-04-29 (Estimated); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Syncytial Virus Infections; Influenza, Human
Keywords: Influenza; Respiratory Syncytial Virus Infections; RSV A Memphis 37
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Influenza, Human

STUDY DESIGN:
Intervention Model Description: GMP influenza A/California/04/2009-like (H1N1); influenza A/Belgium/4217/2015 (H3N2); or RSV Memphis 37 virus strains will be used for experimental infection of volunteers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RSV A Memphis 37 (Experimental): Participants will be inoculated with RSV Memphis 37 virus.
  Interventions: Biological: RSV A Memphis 37
- Influenza A/California/04/2009-like (H1N1) (Experimental): Participants will be inoculated with Influenza A/California/04/2009-like (H1N1).
  Interventions: Biological: Influenza A/California/04/2009-likw (H1N1)
- Influenza A/Belgium/4217/2015 (H3N2) (Experimental): Participants will be inoculated with Influenza A/Belgium/4217/2015 (H3N2).
  Interventions: Biological: Influenza A/Belgium/4217/2015 (H3N2)

INTERVENTIONS:
Biological: RSV A Memphis 37 — Good Manufacturing Practices-certified RSV Memphis 37 10(4) PFU in 1 mL 25% sucrose/DMEM delivered by intranasal drops
  Arms: RSV A Memphis 37
Biological: Influenza A/California/04/2009-likw (H1N1) — Good Manufacturing Practices-certified Influenza A/California/04/09 3.5x10^6 TCID50 in 1 mL in DPBS delivered by intranasal drops
  Arms: Influenza A/California/04/2009-like (H1N1)
Biological: Influenza A/Belgium/4217/2015 (H3N2) — Good Manufacturing Practices-certified Influenza A/Belgium/4217/2015 (H3N2) 3.5x10^6 TCID50 in 1 mL in DPBS delivered by intranasal drops
  Arms: Influenza A/Belgium/4217/2015 (H3N2)

SUMMARY:
Respiratory viruses including influenza and respiratory syncytial virus (RSV) are among the most important causes of severe disease globally, infecting everyone repeatedly throughout life. Understanding of how to prevent infection is incomplete but boosting immunity with vaccines remains the best strategy. T cells have been shown in animals to be essential for clearing respiratory viral infection and are likely to be helpful if stimulated by vaccines. However, where these cells originate from and how they develop in the human lung are still unclear. The investigators will inoculate volunteers with influenza or RSV to examine the relationship between T cells in their blood and lungs and the outcome of infection. By tracking these specialised cells, the investigators aim to develop a better understanding of how they are generated in order to harness them with future vaccines.

DETAILED DESCRIPTION:
Influenza and Respiratory Syncytial Virus (RSV) are the two most common causes of severe viral respiratory tract infection. Seasonal influenza has an overall incidence of 10-20% per annum with frequent complications, and the annual mortality in the USA has been estimated at up to 9.9 deaths per 100,000. According to World Health Organization (WHO) estimates, RSV causes around 64 million infections per annum and 160,000 deaths. It is the leading cause of severe respiratory illness in young children (associated with severe infant wheezing illness) and is also a significant problem in susceptible adults (including the elderly and those with airways disease) in whom RSV is responsible for around 22% of winter respiratory illnesses with a case fatality rate of 2-8%. No vaccines or specific antivirals are available for RSV and those licensed for influenza remain suboptimal. Further understanding of the human immune response to these viruses particularly in the context of the respiratory tract is therefore essential. Experimental human infection studies have the advantage of studying these pathogens in their natural host with the capacity to sample different anatomical sites intensively. Thus the investigators aim to use these models in helping to test vaccines and therapeutics as well as providing critical information on immunity and pathogenesis.

The investigators will use previously characterised Good Manufacturing Practices-certified RSV and influenza viruses derived from recent clinical isolates to investigate the response to infection in healthy adult volunteers. Subjects will be recruited via advertisement and screened at Imperial College London. Healthy individuals will be enrolled in the study and undergo baseline investigations including sampling from blood, upper and lower respiratory tract. They will then be inoculated with RSV or influenza by intranasal drops and quarantined for 10 days. During this time, they will have further blood and respiratory sampling. After the 10 day isolation period, they will be discharged and followed up for up to 6 months post-infection.

These samples will undergo analysis for antibody, B and T cell responses to correlate with outcome of inoculation, which may include no infection, asymptomatic or symptomatic infection. Thus the investigators will infer the role of immune correlates in protection against infection or symptomatic disease.

ELIGIBILITY:
Inclusion Criteria:

- Healthy persons aged 18 to 55 years, able to give informed consent

Exclusion Criteria:

* Chronic respiratory disease (asthma, chronic obstructive pulmonary disease, rhinitis, sinusitis) in adulthood
* Inhaled bronchodilator or steroid use within the last 12 months
* Use of any medication or other product (prescription or over-the-counter) for symptoms of rhinitis or nasal congestion within the last 3 months
* Acute upper respiratory infection (URI or sinusitis) in the past 6 weeks
* Smoking in the past 6 months OR >5 pack-year lifetime history
* Subjects with allergic symptoms present at baseline
* Clinically relevant abnormality on chest X-ray
* Any ECG abnormality
* Those in close domestic contact (i.e. sharing a household with, caring for, or daily face to face contact) with children under 3 years, the elderly (>65 years), immunosuppressed persons, or those with chronic respiratory disease
* Subjects with known or suspected immune deficiency
* Receipt of systemic glucocorticoids (in a dose ≥ 5 mg prednisone daily or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within 6 months prior to challenge
* Known immunoglobulin A deficiency, immotile cilia syndrome, or Kartagener's syndrome
* History of frequent nose bleeds
* Any significant medical condition or prescribed drug deemed by the study doctor to make the participant unsuitable for the study
* Pregnant or breastfeeding women
* Positive urine drug screen
* Detectable baseline haemagglutination inhibition titres against influenza challenge strains
* Influenza arm only: history of hypersensitivity to eggs, egg proteins, gentamicin, gelatin or arginine, or with life-threatening reactions to previous influenza vaccinations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiu, BMBCh PhD, Principal Investigator — Imperial College London
Locations (1):
- National Heart and Lung Institute, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jozwik A, Habibi MS, Paras A, Zhu J, Guvenel A, Dhariwal J, Almond M, Wong EHC, Sykes A, Maybeno M, Del Rosario J, Trujillo-Torralbo MB, Mallia P, Sidney J, Peters B, Kon OM, Sette A, Johnston SL, Openshaw PJ, Chiu C. RSV-specific airway resident memory CD8+ T cells and differential disease severity after experimental human infection. Nat Commun. 2015 Dec 21;6:10224. doi: 10.1038/ncomms10224. PMID 26687547
- [Result] Currie SM, Gwyer Findlay E, McFarlane AJ, Fitch PM, Bottcher B, Colegrave N, Paras A, Jozwik A, Chiu C, Schwarze J, Davidson DJ. Cathelicidins Have Direct Antiviral Activity against Respiratory Syncytial Virus In Vitro and Protective Function In Vivo in Mice and Humans. J Immunol. 2016 Mar 15;196(6):2699-710. doi: 10.4049/jimmunol.1502478. Epub 2016 Feb 12. PMID 26873992
- [Derived] Paterson S, Kar S, Ung SK, Gardener Z, Bergstrom E, Ascough S, Kalyan M, Zyla J, Maertzdorf J, Mollenkopf HJ, Weiner J, Jozwik A, Jarvis H, Jha A, Nicholson BP, Veldman T, Woods CW, Mallia P, Kon OM, Kaufmann SHE, Openshaw PJ, Chiu C. Innate-like Gene Expression of Lung-Resident Memory CD8+ T Cells during Experimental Human Influenza: A Clinical Study. Am J Respir Crit Care Med. 2021 Oct 1;204(7):826-841. doi: 10.1164/rccm.202103-0620OC. PMID 34256007
- [Derived] Guvenel A, Jozwik A, Ascough S, Ung SK, Paterson S, Kalyan M, Gardener Z, Bergstrom E, Kar S, Habibi MS, Paras A, Zhu J, Park M, Dhariwal J, Almond M, Wong EH, Sykes A, Del Rosario J, Trujillo-Torralbo MB, Mallia P, Sidney J, Peters B, Kon OM, Sette A, Johnston SL, Openshaw PJ, Chiu C. Epitope-specific airway-resident CD4+ T cell dynamics during experimental human RSV infection. J Clin Invest. 2020 Jan 2;130(1):523-538. doi: 10.1172/JCI131696. PMID 31815739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RSV A Memphis 37 | Influenza A/California/04/2009-like (H1N1) | Influenza A/Belgium/4217/2015 (H3N2)
Started | 41 | 24 | 10
Completed | 41 | 24 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy adults aged 18-55 years, willing and able to give informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV A Memphis 37 | Influenza A/California/04/2009-like (H1N1) | Influenza A/Belgium/4217/2015 (H3N2) | Total
Number analyzed (Participants) | 41 | 24 | 10 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 24 | 10 | 75
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 26.2 [18 to 52] | 45.3 [22 to 55] | 37.2 [20 to 52] | 33.8 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 5 | 23
  Male | 29 | 18 | 5 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 0 | 11 | 8 | 19
  Asian or Asian British (other) | 0 | 0 | 1 | 1
  White (other) | 0 | 2 | 1 | 3
  Asian or Asian British (Pakistan) | 0 | 0 | 0 | 0
  Mixed (White & Caribbean) | 0 | 1 | 0 | 1
  All other ethnic groups | 0 | 2 | 0 | 2
  White Irish | 0 | 1 | 0 | 1
  Black or Black British (Caribbean) | 0 | 1 | 0 | 1
  Asian or Asian British (Indian) | 0 | 2 | 0 | 2
  Black or Black British (African) | 0 | 3 | 0 | 3
  Unknown | 41 | 0 | 0 | 41
  Mixed White (White & Asian) | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 41 | 24 | 10 | 75

OUTCOME MEASURES:

1. Primary Outcome: Total Symptom Score
Description: Total Symptom Score in infected versus uninfected participants by Jackson's criteria.
  Eight symptoms were evaluated in the symptom diary: nasal discharge, nasal congestion, sneezing, cough, sore throat, headache, feverishness and fatigue. Subjects were asked to score each symptom 0 (absent), 1 (mild), 2 (moderate), 3 (severe). A clinical cold was defined as 2 out of 3 of: a cumulative 14-day symptom score of ≥14; a subjective feeling of a cold; nasal discharge for ≥3 days. Symptoms were evaluated over a longer period than in Jackson's original description to account for an anticipated slower onset and longer duration of illness with RSV compared with rhinovirus. Maximum cumulative symptom score is therefore 336.
Time Frame: 14 days
Population: Total number of participants challenged with the specified challenge virus. For the H1N1 arm, only 22 out of 24 participants were analysed because one participant lost their symptom diary and another was excluded from analysis as they had RSV co-infection
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | RSV A Memphis 37 | Influenza A/California/04/2009-like (H1N1) | Influenza A/Belgium/4217/2015 (H3N2)
Number analyzed (Participants) | 41 | 22 | 10
score on a scale
  Infected: number analyzed (Participants) | 20 | 12 | 7
  Infected | 29.25 [8.50 to 47.50] | 17.50 [8.75 to 23.00] | 11.00 [7.50 to 18.75]
  Uninfected: number analyzed (Participants) | 21 | 10 | 3
  Uninfected | 13.00 [4.75 to 22.00] | 0 [0 to 1.25] | 1 [0 to 4]

2. Secondary Outcome: Frequency of T Cells in Blood by Flow Cytometry
Description: Peak Ki-67+ CD38+ CD8+ T cells in the blood by flow cytometry.
Time Frame: 6 months
Population: For the H1N1 arm, one participant was excluded from analysis as they had RSV co-infection.
  For the RSV arm, only 32/41 participants were analysed because there were insufficient PBMCs from the remaining participants to run the analysis
Measure: Median (Inter-Quartile Range); unit: % of CD8+ lymphocytes
Arm/Group | RSV A Memphis 37 | Influenza A/California/04/2009-like (H1N1) | Influenza A/Belgium/4217/2015 (H3N2)
Number analyzed (Participants) | 32 | 23 | 7
% of CD8+ lymphocytes
  Infected: number analyzed (Participants) | 17 | 13 | 4
  Infected | 0.79 [0.42 to 1.10] | 3.81 [2.46 to 5.56] | 4.13 [2.55 to 16.21]
  Uninfected: number analyzed (Participants) | 15 | 10 | 3
  Uninfected | 0.49 [0.24 to 0.81] | 0.985 [0.752 to 1.535] | 1.18 [0.77 to 1.59]

3. Secondary Outcome: Frequency of T Cells in Respiratory Tract by Flow Cytometry
Description: Peak Ki-67+ CD38+ CD8+ T cells in bronchoalveolar lavage (BAL) by flow cytometry
Time Frame: 6 months
Population: For the H1N1 arm, one participant was excluded from analysis as they had RSV co-infection.
  For the RSV arm, only 20/41 participants were analysed because there were insufficient airway cells from some participants to run the analysis.
  For the H3N2 arm, the analysis was not run on the 3 uninfected participants. Only 3 were analysed in the infected participants because 1 participant was excluded for co-infection and the other 3 participants had insufficient airway cells to run the analysis.
Measure: Median (Inter-Quartile Range); unit: % of CD8+ lymphocytes
Arm/Group | RSV A Memphis 37 | Influenza A/California/04/2009-like (H1N1) | Influenza A/Belgium/4217/2015 (H3N2)
Number analyzed (Participants) | 20 | 23 | 3
% of CD8+ lymphocytes
  Infected: number analyzed (Participants) | 10 | 13 | 3
  Infected | 2.21 [0.96 to 3.80] | 81.15 [0 to 90.48] | 4.36 [1.35 to 5.49]
  Uninfected: number analyzed (Participants) | 10 | 10 | 0
  Uninfected | 0.65 [0.27 to 1.11] | 0.412 [0.187 to 0.598] |

4. Secondary Outcome: Viral Load
Description: Nasal wash viral load by quantitative polymerase chain reaction (qPCR) (Area under curve)
Time Frame: 28 days
Population: For the H1N1 arm, one participant was excluded from analysis as they had RSV co-infection.
Measure: Median (Inter-Quartile Range); unit: log10 copies*days/mL
Arm/Group | RSV A Memphis 37 | Influenza A/California/04/2009-like (H1N1) | Influenza A/Belgium/4217/2015 (H3N2)
Number analyzed (Participants) | 41 | 23 | 10
log10 copies*days/mL
  Infected: number analyzed (Participants) | 20 | 13 | 7
  Infected | 18.24 [11.51 to 24.34] | 5.85 [0.82 to 9.22] | 26.40 [5.52 to 33.13]
  Uninfected: number analyzed (Participants) | 21 | 10 | 3
  Uninfected | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Frequency of T Cells in Blood by Enzyme-linked Immunospot (ELISpot)
Description: Peak T cells in blood by Enzyme-linked Immunospot (ELISpot). IFNy SFU/million PBMCs (Spot Forming Unit)
Time Frame: 6 months
Population: For the H1N1 arm, there were only enough remaining PBMCs from 14 participants. For the H3N2 arm, there were insufficient cells to run the analysis. For the RSV arm, only 18/41 participants were analysed because there were insufficient PBMCs from the remaining participants to run the analysis.
Measure: Median (Inter-Quartile Range); unit: IFNy SFU/million PBMCs
Arm/Group | RSV A Memphis 37 | Influenza A/California/04/2009-like (H1N1) | Influenza A/Belgium/4217/2015 (H3N2)
Number analyzed (Participants) | 18 | 14 | 0
IFNy SFU/million PBMCs
  Infected: number analyzed (Participants) | 10 | 8 | 0
  Infected | 778.30 [459.20 to 1228] | 161 [128 to 214] |
  Uninfected: number analyzed (Participants) | 8 | 6 | 0
  Uninfected | 159.20 [43.75 to 419.2] | 29 [21 to 43] |

ADVERSE EVENTS:
Time Frame: Through study completion, average 6 months
Description: Subjects may experience symptoms of a common cold which would not be deemed AEs.
  A fever >38ºC for >3 consecutive days or withdrawal due to intolerable symptoms in >2 subjects will lead to study suspension. A DSMB will be determine any systematic cause for unexpectedly severe symptoms.
  Any influenza-like illness resulting in Sustained elevated HR >120bpm AND Sustained low SBP <100 Sustained elevated RR >30/min AND Sustained low O2 sats <94% Evidence of pneumonia New ECG abnormalities
Arm/Group | RSV A Memphis 37 | Influenza A/California/04/2009-like (H1N1) | Influenza A/Belgium/4217/2015 (H3N2)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/24 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/24 | 0/10
Other Adverse Events (participants affected / at risk) | 0/41 | 0/24 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT02755948/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT02755948/ICF_001.pdf